CLINICAL TRIAL: NCT02362789
Title: Exploratory Study on the Kinetics of Psoriasis Symptoms, Pruritus Intensity and Lesional Biomarkers in Patients With Moderate to Severe Plaque-type Psoriasis Treated With Subcutaneous Secukinumab (300 mg) During a 16 Week Open-label run-in Phase Followed by a 16 Week Randomized, Double-blind, Placebo-controlled Withdrawal Phase
Brief Title: Secukinumab Study in PSOriasis Exploring pruRITUS Intensity and Lesional Biomarkers
Acronym: PSORITUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457ADE03
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secukinumab (Experimental): 300 mg secukinumab (administered as two injections of 150 mg each) at Weeks 16, 20, 24, and 28
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Inactive ingredients administered as a matching placebo at Weeks 16, 20, 24, and 28
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab — 150 mg secukinumab in 1 ml solution for subcutaneous injection (pre-filled syringe)
  Arms: Secukinumab
Biological: Placebo — Matching placebo in 1 ml solution for subcutaneous injection (pre-filled syringe)
  Arms: Placebo

SUMMARY:
The study is designed to explore the kinetics of psoriasis symptoms, pruritus intensity and lesional biomarkers.

DETAILED DESCRIPTION:
All subjects will undergo a 16 week run-in phase (open label). At Week 16, an evaluation of the PASI response will be performed. Patients who achieve a PASI reduction of less than 98 percent will complete the study at Week 16 and be referred to routine clinical care for psoriasis by the investigator. Patients who achieve extensive remission (PASI reduction by 98-100 percent) at Week 16 will enter the randomized withdrawal phase (blinded) where they will be randomized to receive either secukinumab or matching placebo and will complete the study at Week 32.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic moderate to severe plaque type psoriasis as diagnosed by a qualified physician at least 6 months prior to baseline and with a PASI score > 10 at baseline.
* Psoriasis patients with pruritus intensity of ≥ 30 on a 100-point VAS, with a recall period of 24h as part of the PGA-CP, both, at screening and at baseline.

Key Exclusion Criteria:

* Underlying conditions other than psoriasis which in the opinion of the investigator currently cause or influence pruritus of the skin (e.g. drug induced pruritus, renal insufficiency, diabetes).
* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic, and guttate) at screening or study start.
* Ongoing use of prohibited psoriasis and non-psoriasis treatments. Washout periods have to be adhered to. If the use of any of the prohibited treatments is required, then the subject may not be included into the study.
* Pregnancy, breast feeding or inadequate contraception (if necessary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-01-04 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Lead, Principal Investigator — Muenster
Locations (18):
- Germany (18):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dippoldiswalde-Schmiedeberg
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Selters
  - Novartis Investigative Site, Stuttgart

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 132 subjects enrolled in the study, 130 entered the Run-In phase.
Groups:
- Run-in: 300 mg secukinumab (administered as two injections of 150 mg each) at Weeks 0, 1, 2, 3, 4, 8, and 12
Period: Run-in Phase (Week 0 to 16)
Arm/Group | Run-in | Secukinumab | Placebo
Started | 130 | 0 | 0
Completed | 128 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Death unrelated to study treatment | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Randomized Withdrawal (Wk 16 to 32)
Arm/Group | Run-in | Secukinumab | Placebo
Started | 0 (N/A. Run-in phase completed.) | 42 (Subjects achieving PASI reduction by 98-100% vs. baseline during Run-In) | 38 (Subjects achieving PASI reduction by 98-100% vs. baseline during Run-In)
Completed | 0 | 38 | 26
Not Completed | 0 | 4 | 12
Not completed — Lack of Efficacy | 0 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 4
Not completed — Subject/guardian decision | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (randomized withdrawal phase) (FAS-R). All patients that received at least one dose of blinded study drug during the randomized withdrawal phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Customized [Count of Participants; unit: Participants]
  <65 | 37 | 36 | 73
  >=65 | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 27 | 22 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 41 | 0 | 41
  Black | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pruritus Intensity Visual Analogue Scale Score at Week 32
Description: On a 100-mm horizontal line, the patient placed a mark representing their perception of worst itching (pruritus) within a recall period of 24 hours, where 0 = no pruritus and 100 = most severe pruritus.
Time Frame: Week 32
Population: FAS-R, LOCF
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 42 | 38
Units on a scale | 8.8 (4.7) | 27.1 (4.9)
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Test type: Superiority; p = 0.0055, ANCOVA; Mean Difference (Net) = -18.3, 95% CI 2-sided [-31.01 to -5.59]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 1 year, 3 months.
Description: The safety set included all patients that received at least one dose of study drug.
Arm/Group | Run-In | Secukinumab | Placebo
Serious Adverse Events (participants affected / at risk) | 6/130 | 2/42 | 0/38
Other Adverse Events (participants affected / at risk) | 43/130 | 16/42 | 19/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In (N=130) | Secukinumab (N=42) | Placebo (N=38)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANEURYSM RUPTURED (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In (N=130) | Secukinumab (N=42) | Placebo (N=38)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 3
INFLUENZA (Infections and infestations) | 2 | 1 | 2
NASOPHARYNGITIS (Infections and infestations) | 31 | 12 | 11
RHINITIS (Infections and infestations) | 0 | 1 | 2
SINUSITIS (Infections and infestations) | 0 | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 0 | 0
HEADACHE (Nervous system disorders) | 5 | 3 | 1
HYPERTENSION (Vascular disorders) | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.